CLINICAL TRIAL: NCT00003850
Title: A Phase II Study of Thalidomide in Recurrent and Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Thalidomide in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02299; MDA-ID-98270; NCI-T98-0074; CDR0000067011 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2001-01

CONDITIONS: Head and Neck Cancer
Keywords: recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Thalidomide

ARMS (1):
- Arm I (Experimental): Patients receive 4-20 capsules of oral thalidomide once daily. Dose is escalated in individual patients on a weekly basis for the first 5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity, or for 12 months past complete response.
  Interventions: Drug: thalidomide

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
Phase II trial to study the effectiveness of thalidomide in treating patients with recurrent or metastatic head and neck cancer. Thalidomide may stop the growth of head and neck cancer by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the effect of thalidomide on survival of patients with recurrent or metastatic squamous cell carcinoma of the head and neck.

II. Determine clinical response rates following this therapy in these patients. III. Determine the toxic effects of thalidomide in these patients. IV. Determine the effect of thalidomide on tumor angiogenesis in these patients.

OUTLINE:

Patients receive 4-20 capsules of oral thalidomide once daily. Dose is escalated in individual patients on a weekly basis for the first 5 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity, or for 12 months past complete response.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven squamous cell carcinoma of the head and neck
* Recurrent disease OR metastatic disease at initial diagnosis or at recurrence
* Initial therapy of surgery and/or radiotherapy, induction chemotherapy, or concurrent chemotherapy and radiotherapy allowed
* No more than one prior regimen of chemotherapy or biologic therapy for metastatic disease
* Recurrence after adjuvant or induction chemotherapy may have received one additional course of chemotherapy or biologic therapy

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: Zubrod 0-2
* Life expectancy: At least 3 months
* WBC at least 3000/mm3
* Platelet count at least 100,000/mm3
* Hematocrit at least 30%
* Bilirubin no greater than 1.5 times normal
* SGOT/SGPT no greater than 1.5 times normal
* Creatinine no greater than 1.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile women must use 2 methods of effective contraception, 1 barrier and 1 hormonal, beginning at least 4 weeks before study and continuing during and for 1 month after study
* Men must use effective barrier contraception during and for 1 month after study
* No grade 2 or greater peripheral neuropathy
* No serious infection or other concurrent illness requiring immediate therapy
* Must be able to take oral medications
* No medical or social factors that would interfere with compliance

PRIOR CONCURRENT THERAPY:

* Any number of courses of one regimen of chemotherapy allowed
* No concurrent cytotoxic chemotherapy
* No concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 1999-04; Primary Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy S. Herbst, MD, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States